CLINICAL TRIAL: NCT03056950
Title: BFR DISTRAD NON OP: Blood Flow Restricted Training During Rehabilitation Following Distal Radius Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jill Cancio, Principal Investigator, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C.2016.045
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Distal Radius Fracture; Rehabilitation
Keywords: Blood Flow Restriciton; Occlusion training; Distal radius fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non-oclusion training group (No Intervention): The control (non-occlusion training) group will follow the standard s/p distal radius fracture rehabilitation protocol. Treatment will include passive, active assistive,active range of motion (P/AA/AROM) to wrist, forearm and hand; desensitization as needed; edema control as needed; heat/cold modalities as needed; and strengthening exercises.
- occlusion traingn with tourniquet (Active Comparator): The occlusion training group will follow the same protocol as described above but will utilize occlusion training with the strengthening exercises. Investigators will use an established occlusion training protocol already being used. Intervention: Occlusion training with tourniquet (DELFI PTS ii portable tourniquet system)
  Interventions: Device: DELFI PTS ii portable tourniquet

INTERVENTIONS:
Device: DELFI PTS ii portable tourniquet — A cuff will be wrapped around the most proximal portion of the arm of the involved extremity. In order to individualize the pressure for each subject, the limb occlusion pressure will be measured (with doppler ultrasound over the radial artery at the wrist level) at the first scheduled therapy visit. The cuff pressure utilized during the post-operative exercises will be set at 50% of the limb occlusion pressure. The subjects' strength will be re-assessed approximately every 2-4 weeks and the load will be increased as tolerated.
  Arms: occlusion traingn with tourniquet

SUMMARY:
Occlusion training, resistance exercise performed with a specialized venous tourniquet, leads to beneficial changes in muscle strength at low resistance and minimal stress on the nearby joint. This novel resistance training has the potential to greatly improve muscle strength gains in individuals who are unable, for medical reasons, to perform the high resistance exercises typically required to improve strength. Our study will examine the effect of this technique on strength recovery following distal radius fracture treated with cast immobilization (non-operatively). The primary objective of the intervention is to achieve accelerated recovery of forearm, wrist and hand function as assessed using measures such as grip/pinch strength, validated questionnaires, and functional outcome testing. Occlusion training can potentially serve as a specialty intervention for rehabilitation patients, reduce the cost of care, and improve the treatment options for both patients and providers.

DETAILED DESCRIPTION:
Investigator's will perform a prospective, randomized, controlled study. All subjects in this group will be adults who have sustained a distal radius fractured treated with cast immobilization (non-operative) at San Antonio Military Medical Center (SAMMC) clinic system. Participants will be provided information about the study and inclusion/exclusion criteria, and upon conclusion of the formal consenting process, and signature of the consent document, will be considered enrolled in the study. Prior to intiation of any study procedures each patient must be cleared for participation in treatment by his or her surgeon as per standard post-fracture protocol. Medical clearance will be documented on the Enrollment form (Appendix A) and the Medical History form (Appendix K). This will be verified by accessing the medical record to confirm that a referral was made for post-fracture rehabilitation. Before initiation of treatment, the enrolled subjects will be randomized to either a standard rehabilitation group or an occlusion training rehabilitation group. Randomization with be performed with a random number generator. Treatment will be initiated approxmiately 6 weeks s/p fracture (when cleared by the orthopedic surgeon). Participantswill undergo approximetely 8-12 weeks of treatment with therapy sessions two to three days a week (consistent with standard of care), and will have re-assessments completed at approximately 4 weeks, 8 weeks, and 12 weeks after initiating the training protocol. The 12-week time point (after initiation of therapy) will be at approximately the same time that patients are released for full activity per standard of care.

The control (non-occlusion training) group will follow the standard s/p distal radius fracture rehabilitation protocol. Treatment will include passive, active assistive,active range of motion (P/AA/AROM) to wrist, forearm and hand; desensitization as needed; edema control as needed; heat/cold modalities as needed; and strengthening exercises. Specific strengthening exercises will include wrist flexion/extension over a foam wedge, forearm pronation/supination with arm positioned at side and elbow at 90 degrees, thumb opposition (pinch strength) as well as grip strengthening. The amount of resistance used with be determined by patient tolerance and post operative precautions.

The occlusion training group will follow the same protocol as described above but will utilize occlusion training with the strengthening exercises. We will use an established occlusion training protocol already being used at the CFI. The resistance for strength training will be determined based on the individual participants tolerance. A cuff will be wrapped around the most proximal portion of the arm of the involved extremity. In order to individualize the pressure for each subject, the limb occlusion pressure will be measured (with dopplar ultrasound over the radial artery at the wrist level) at the first scheduled therapy visit. Limb occlusion pressure is the pressure necessary to completely occlude arterial blood flow. The cuff pressure utilized during the post-operative exercises will be set at 50% of the limb occlusion pressure. Repetions will be 30, 15, 15 and 15 for each of the four sets. A 30-second rest will be given between sets. The tourniquet will stay inflated throughout the entire exercise and rest sessions, and no longer than 30 minutes consecutively for any time that the tourniquet is inflated. After completion of the 4 sets the tourniquet pressure will be deflated. The subjects' strength will be re-assessed approximately every 2-4 weeks and the load will be increased as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Status post distal radius fracture (non-operative treated with cast immobilization)
* Males and females 18-65 years of age
* Eligible to receive care at Military Treatment Facility (DEERS eligible)
* Must be able to read and write in English in order to consent

Exclusion Criteria:

* Contralateral upper extremity involvement resulting in less than normal range of motion, muscle strength, or daily pain greater than 1/10.
* Status post distal radius fractured treated operatively (k-wires, ORIF, etc)
* Pregnancy - per patient self-report. Due the expected small number of pregnant individuals and resulting inability to account for its effect on resulting outcomes, these patients will not be included in the study.
* Recent history of deep vein thrombosis, within the 12 months or on active treatment with anticoagulants
* History of upper quadrant lymph node dissection
* History of endothelial dysfunction
* Patient endorsement of easy bruising
* Active Infection in the injured arm
* Cancer (current diagnosis per medical record)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
grip strength | 18 weeks
  grip strength will be assessed using the JAMAR Hand Dynamometer

SECONDARY OUTCOMES:
pinch strength | 18 weeks
  Pinch strength will be assessed using the PG-60 Pinch Gauge. The mean of three successive trials will be recorded for each pinch position (tip, key and palmar)
joint range of motion | 18 weeks
  Joint range of motion (ROM) will be assessed using a plastic goniometer

OTHER OUTCOMES:
Performance measure DASH | 18 weeks
  a 30-item self-report measure that assesses a subject's perceived ability to complete twenty-one upper extremity functional activities using a 5-point Likert scale. The cumulative DASH score is scaled from 0 to 100, with higher scores indicating increased disability
Performance measure PRWE | 18 weeks
  a 15-item questionnaire that assesses wrist pain (5 items) and disability (10 items) in activities of daily living.
Performance measure JTHFT | 18 weeks
  is a seven part test that evaluates the time needed to perform seven hand-related tasks
Performance measure PSFS | 18 weeks
  a patient-specific outcome measure to assess functional status[49]. The patient is asked to identify three to five activities that he or she has difficulty performing due to his or her condition. The patient then rates the amount of limitation he or she has in performing each of these activities on an 11-point scale with 0 being unable to perform the activity and 10 being able to perform the activity with no problem. An average score for the activities gives an ability score out of 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided